CLINICAL TRIAL: NCT04382417
Title: Characteristics and Outcomes of Critically Ill Patients With Covid-19 in a Large Swedish County Hospital - a Prospective Observational Cohort Study
Brief Title: Prospective Observational Cohort Study of Critically Ill Patients With Covid-19 in Sweden
Status: Completed | Type: Observational
Sponsor: Region Västmanland (Other)
Responsible Party: Principal Investigator, Erland Ostberg, M.D., Ph.D., Region Västmanland
Other Study IDs: RegionVastmanland
Record Dates: First submitted 2020-05-04; First posted 2020-05-11 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Covid-19; Critical Illness
MeSH Terms: conditions — COVID-19; Critical Illness | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid-19: Patients with verified or highly suggestive Covid-19 diagnosis and Intensive Care treatment.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Not required

SUMMARY:
The study will prospectively collect data from patients with Covid-19 admitted to the Västerås Intensive Care Unit, Västerås Hospital. Demographic, clinical, radiographic and laboratory characteristics will be recorded. Analysis of data to identify predictors of disease severity, mortality and treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Intensive Care Unit with biological samples positive for SARS-CoV-2.
* Patients admitted to the Intensive Care Unit with one or more negative tests but with clinical and radiological characteristics highly suggestive of SARS-CoV-2 and thus considered positive for the disease.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Covid-19.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2020-03-26 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | At 90 days follow-up after admittance to Intensive Care

SECONDARY OUTCOMES:
Hospital length of stay | Until 90 days after admittance to Intensive Care
ICU length of stay | Until 90 days after admittance to Intensive Care
Number of days on mechanical ventilation | Until 90 days after admittance to Intensive Care
Number of patients receiving vasopressor support | Until 90 days after admittance to Intensive Care
Number of patients receiving renal replacement therapy | Until 90 days after admittance to Intensive Care
Patient characteristics | At admission to ICU

CONTACTS AND LOCATIONS:
Overall Officials: Erland Östberg, M.D., Ph.D., Principal Investigator — Region Västmanland
Locations (1):
- Intensive Care Unit, Västerås Hospital, Västerås, Västmanland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided